CLINICAL TRIAL: NCT07372872
Title: Development and Feasibility Testing of the "MyGlucoCare" Smartphone-Based Self-Management for Personalised Support of Women With Gestational Diabetes
Brief Title: Feasibility Testing of the "MyGlucoCare" Smartphone App for Women With Gestational Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Bronya LUK Hi Kwan, Assistant Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PFDS/2025/21; PFDS/2025/21 (Other Grant/Funding Number: Hong Kong Metropolitan University)
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: GDM; Smartphone-Based Self-Management; Personalised Support
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "MyGlucoCare" intervention (Experimental): The "MyGlucoCare" intervention is a comprehensive, technology-facilitated program delivered over 8 to 12 weeks.
  Interventions: Device: MyGlucoCare

INTERVENTIONS:
Device: MyGlucoCare — The "MyGlucoCare" intervention is a comprehensive, technology-facilitated program delivered over 8 to 12 weeks. It integrates three core components to provide holistic and personalised support for women with gestational diabetes (GDM).

SUMMARY:
The goal of this pilot study is to test the feasibility and preliminary impact of "MyGlucoCare," a smartphone-based program designed to support women with gestational diabetes (GDM). The main questions it aims to answer are:

Is the "MyGlucoCare" program practical and acceptable for participants?

Does it show preliminary signs of improving self-management, blood sugar control, and well-being in women with gestational diabetes (GDM)?

Researchers will conduct a single-arm study to gather initial data on the program's use and effects, which will be used to plan a larger future clinical trial.

Participants will:

Use the "MyGlucoCare" app for 8-12 weeks during their pregnancy.

Receive personalized education, support from a clinician, and access to a moderated peer group through the app.

Complete questionnaires and log health data via the app at the start, near the end of pregnancy, and after giving birth.

Some participants will also take part in an interview to share their feedback on the program.

DETAILED DESCRIPTION:
1. Project Objectives

   The objective of this pilot study is to evaluate the feasibility, acceptability, and preliminary impact of the "MyGlucoCare" smartphone program, which provides holistic self-management support for women with gestational diabetes mellitus (GDM).

   The primary aim is to determine the feasibility of the research procedures and the acceptability of the "MyGlucoCare" program itself. This will involve assessing participant recruitment, retention, and data completion rates to evaluate feasibility. The program's acceptability and usability will be evaluated from the participants' perspective by measuring their engagement and subjective experiences.

   The secondary aim is to gather preliminary evidence of the program's potential impact. This includes obtaining initial estimates of its effect on self-efficacy for diabetes management and self-reported self-management behaviours. The study will also explore preliminary changes in key clinical and behavioural markers, specifically glycemic control (measured by pre- and post-meal blood glucose levels), physical activity levels, and perceived stress levels. Finally, a descriptive exploration of relevant maternal and neonatal pregnancy outcomes will be conducted to inform future research.
2. Project Plan and Methodology

   Study Design: A single-arm pilot study with a pre-test/post-test design.

   Sample Size A pragmatic sample of 30 women will be recruited. This sample size is consistent with recommendations for pilot studies to obtain reliable estimates of feasibility parameters and is not intended for formal hypothesis testing.

   Recruitment Strategy A multi-faceted strategy will ensure timely participant enrolment. This will consist of community-based recruitment using targeted advertisements on Hong Kong parenting forums and social media, supplemented by snowball sampling.

   Eligibility Criteria Eligible participants will be pregnant women diagnosed with GDM via a 75g Oral Glucose Tolerance Test (OGTT), conducted between 24 and 28 weeks of gestation. Participants must be aged 18 years or older, own a smartphone with reliable internet access, and be able to read and understand Chinese.

   Potential participants will be excluded from the study if they have a pre-existing diagnosis of Type 1 or Type 2 diabetes mellitus, a known major fetal anomaly, or are concurrently enrolled in any other structured GDM self-management intervention. Individuals with severe mental health conditions that could impair their ability to use the technology-based intervention will also be excluded.

   The "MyGlucoCare" Intervention The "MyGlucoCare" intervention is a comprehensive, technology-facilitated program delivered over 8 to 12 weeks. It integrates three core components to provide holistic and personalised support for women with GDM.

   Component A: Personalised Education & Skill-Building (Automated) This component delivers a structured curriculum through automated messages and posts within the MyGlucoCare platform. The educational content covers essential topics for gestational diabetes (GDM) management, including disease education, dietary guidance using food exchange tables, safe exercise routines, stress management techniques, community resource information, advice for dining out, supporting services for pregnant mothers, and postpartum planning information encompassing breastfeeding and newborn care.

   Component B: Proactive Personalised Support (Driven by Clinicians) A dedicated study nurse or midwife provides individualised clinical support through the MyGlucoCare platform. Support is delivered via two primary methods: proactive, scheduled check-ins and responsive communication. The clinician will initiate bi-weekly contact to review glucose logs, identify personal barriers to self-management, and collaboratively set individualised goals. Furthermore, participants can use the platform's chat function to ask questions at any time, receiving a response from the clinician within 24 hours on weekdays.

   Component C: Facilitated Peer Support (Moderated) To foster a sense of community and shared experience, a private peer support group will be established using an integrated chat function. This group will be lightly moderated by the research team to encourage the exchange of experiences and practical tips while maintaining a safe, positive, and supportive environment for all participants.

   Data Collection & Measures Data will be collected at three time points: Baseline (T0), post-intervention (T1, at approximately 36 weeks' gestation), and Postpartum (T2, 6-12 weeks after delivery). Data collection will be facilitated through the MyGlucoCare platform, and participant interviews.

   Feasibility Metrics will be systematically tracked and include screening logs to determine recruitment rates, study completion data to calculate retention rates, adherence to scheduled support calls, and quantitative engagement metrics with the platform's chat features.

   Acceptability & Usability will be assessed using a mixed-methods approach. Quantitatively, the standardized 10-item System Usability Scale (SUS) will be administered. Qualitatively, semi-structured interviews will be conducted with a sub-sample of approximately 10 participants to explore their experiences, the perceived usefulness of the program, and to gather detailed suggestions for improvement.

   Preliminary Outcome Measures will be collected to inform a future definitive trial. These include:
   * Self-Efficacy for Diabetes Management measured using the Diabetes Management Self-Efficacy Scale.
   * Self-Management Behaviours, assessed with a Diabetes Self-Management Questionnaire (SDSCA).
   * Glycaemic Control, evaluated through self-monitored pre-meal and 2-hour post-meal blood glucose levels (between T0 and T1) and the results of a postpartum Oral Glucose Tolerance Test (OGTT) at T2.
   * Psychological Well-being measured using the Patient Health Questionnaire-9 (PHQ-9).
   * Participant-Reported pregnancy outcomes: Maternal and Infant Outcomes, collected from medical records at T2.

   Data Analysis Quantitative Analysis: Descriptive statistics (means, frequencies, standard deviations) will be used for feasibility outcomes and participant characteristics. Pre-post changes in outcome measures will be analysed using paired t-tests or Wilcoxon signed-rank tests, with a focus on estimating effect sizes and confidence intervals for future sample size calculation. Qualitative Analysis: Thematic analysis will be applied to the interview transcripts to identify key themes related to acceptability and suggestions for refinement.

   Ethical Considerations Ethical approval has been obtained from the HKMU Research ethical committee. Written informed consent will be obtained from all participants. All data will be anonymized and stored securely. Confidentiality within the peer group will be emphasized in the group rules.
3. Expected Outputs or Deliverables

This pilot study will generate essential deliverables to support future research and implementation:

1. A Validated "MyGlucoCare" Intervention Protocol: A ready-to-use package including the educational curriculum, clinician support guidelines, and peer moderation framework, refined through user feedback.
2. Feasibility and Acceptability Evidence: A clear report quantifying recruitment, retention, and engagement rates, alongside participant feedback on usability and satisfaction, to determine the viability of a full-scale trial.
3. Preliminary Efficacy Data for RCT Planning: Initial data on changes in self-efficacy, self-management, and glycaemic control will inform the sample size calculation and methodology for a definitive randomized controlled trial. Crucially, these findings will directly address reviewer comments on the submitted FDS proposal (UGC/FDS16/M27/25) regarding the need for pilot data, thereby strengthening the revised application and increasing its chance of success in the next resubmission round.
4. To ensure broad impact, the findings will be actively disseminated. A minimum of one manuscript is planned for submission to high-impact, peer-reviewed journals, such as JMIR Diabetes for primary outcomes on usability and acceptance. Preliminary results will be presented at international conferences, including the East Asian Forum of Nursing Scholars and the International Congress on Midwifery. Furthermore, findings will be shared with local healthcare partners to facilitate translation into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with Gestational Diabetes Mellitus (GDM) via a 75g Oral Glucose Tolerance Test (OGTT), conducted between 24 and 28 weeks of gestation (Hong Kong College of Obstetricians and Gynaecologists, 2016).
* Aged 18 years or older.
* Own a smartphone with reliable internet access.
* Able to read and understand Chinese.

Exclusion Criteria:

* Pre-existing diagnosis of Type 1 or Type 2 diabetes mellitus.
* Known major fetal anomaly.
* Concurrent enrollment in any other structured GDM self-management intervention.
* Severe mental health conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women diagnosed with gestational diabetes (GDM) via a 75g Oral Glucose Tolerance Test (OGTT), conducted between 24 and 28 weeks of gestation
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Enagagement | 8-12 weeks
  Measures participant interaction with the study protocol and app (%). • Measures: Mean/median frequency of (e.g., per week)
Recruitment & Retention Rates | 8-12 weeks
  Assesses the practicality of executing the trial. • Unit of Measure: Proportion/Percentage (%) for each
System Usability | 8-12 weeks
  Quantifies the perceived usability of the "MyGlucoCare" app using a validated instrument.• Measure: Mean score on the System Usability Scale (SUS). • Unit of Measure: Score on a scale (0-100).

SECONDARY OUTCOMES:
Secondary outcome measures | All changes measured from baseline (T0) to post-intervention (T1, 8-12 weeks), except postpartum OGTT and delivery outcomes collected at T2 (postpartum period).
  Change in Diabetes Management Self-Efficacy Score (DMSES, 20-200; higher=better).
  Change in Diabetes Self-Care Activities frequency (SDSCA, 0-7 days/week; higher=better).
  Change in Self-Monitored Blood Glucose (fasting & postprandial mmol/L; lower=better).
  Postpartum Glucose Tolerance Status (% with normal OGTT at 6-12 weeks postpartum).
  Change in Depressive Symptom Score (PHQ-9, 0-27; higher=worse). Maternal and Neonatal Delivery Outcomes: gestational age, mode of delivery, birth weight, and neonatal hypoglycemia.

IPD SHARING:
Plan to Share IPD: No
The study is conducted under ethical approval which, along with the participant consent forms, does not include provisions for public sharing of individual-level data. Sharing IPD would violate the confidentiality agreement with our participants. Aggregated data will be presented in publications.

REFERENCES:
- [Result] Wang, Y., Lei, T., & Liu, X. (2020). Chinese System Usability Scale: Translation, Revision, Psychological Measurement. International Journal of Human-Computer Interaction, 36(10), 953-963. https://doi.org/10.1080/10447318.2019.1700644
- [Result] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Result] Ritter, P. L., Lorig, K., & Laurent, D. D. (2016). Characteristics of the Spanish- and English-Language Self-Efficacy to Manage Diabetes Scales. The Diabetes Educator, 42(2), 167-177. https://doi.org/10.1177/0145721716628648
- [Result] O'Neill, B. (2022). Sample size determination with a pilot study. PLoS ONE, 17(2 February). https://doi.org/10.1371/journal.pone.0262804
- [Result] Lorig, K. R., Ritter, P. L., & González, V. M. (2003). Nursing Research (Vol. 52, Issue 6). http://journals.lww.com/nursingresearchonline
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Hong Kong College of Obstetricians and Gynaecologists. (2016). HKCOG Guidelines Guidelines for the Management of Gestational Diabetes Mellitus.
- [Result] Jordan, P. W., Thomas, B., McClelland, I. L., & Weerdmeester, B. (1996). Usability evaluation in industry. CRC press